CLINICAL TRIAL: NCT07162545
Title: "Effects Of Stroboskobic Visual Training On Cognitive Performance in Adolescent Male Volleyball Players
Brief Title: Effects Of Stroboskobic Visual Training On Cognitive Performance in Adolescent Male Volleyball Players.
Status: Recruiting | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Oguzhan Bahadir DEMIR, Assist. Prof., Kocaeli University
Other Study IDs: Karabuk, 2025/2432
Record Dates: First submitted 2025-08-24; First posted 2025-09-09 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Orientation
Keywords: Attention; Cognition; Reaction Time
MeSH Terms: conditions — Orientation, Spatial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study: Training Program: Stroboscopic visual training program to be applied 2 days a week, for 8 weeks.
  Interventions: Other: stroboskopic visual training
- control: Routine training program

INTERVENTIONS:
Other: stroboskopic visual training — Players in the study group will wear stroboscopic glasses for 10 minutes a day, two days a week, for eight weeks during their routine training. Evaluations will be repeated at the end of the eight weeks.
  Groups: study

SUMMARY:
Objective: To determine the effects of a stroboscopic training program on cognitive function in adolescent male volleyball players. The study aims to reveal the impact of using stroboscopic glasses during a portion of their training on volleyball players' cognitive functions.

The data obtained from the study will be important for improving volleyball training programs and contributing to the sports science literature.

DETAILED DESCRIPTION:
Numerous studies have shown that physical activity produces structural and functional changes in the brain that support cognitive functions. Some studies suggest that different types of exercise have different effects on cognition. A growing body of literature suggests that the effects of physical exercise on cognitive function may be related to the type of exercise.

Sports are divided into two groups based on the predictability and consistency of the performance environment: open and closed skill sports. Open skill sports (e.g., volleyball, tennis, soccer, etc.) are externally paced activities performed in a dynamic, unpredictable environment, while closed skill sports (e.g., running, swimming, archery, etc.) are internally paced and performed in a static, predictable environment. A recent study showed that team athletes outperform recreational athletes in sustained attention and processing speed. Volleyball, as a team sport, may further enhance some aspects of cognitive skills.

The purpose of this study was to examine the effects of volleyball training using stroboscopic glasses on cognitive function in adolescent male volleyball players.

Effects of Stroboscopic Visual Training: Humans have a remarkable capacity for learning and adaptation. The disruption of visual information can force individuals to reduce their reliance on online visual feedback. It is believed that practicing in situations where visual input is poor will force individuals to better utilize the limited visual information available. This can train the perceptual and attentional abilities that support basic visuomotor control. Attention is a critical skill in many domains, and even a small increase can have profound effects; a small improvement in motion perception and focused attention is crucial for a competitive athlete or a soldier searching for an enemy combatant. Perceptual information influences many motor tasks and ensures the maintenance of accurate control in changing or uncertain environments. Consequently, changes in the environment will regularly produce variations in task performance.

ELIGIBILITY:
Inclusion Criteria:

* Being an adolescent male volleyball player between the ages of 13-18.
* Having attended volleyball training regularly for at least one year.
* Agreeing to attend training regularly throughout the study period.
* Having signed the voluntary participation form and parental consent form.
* Having no visual or auditory impairments.
* Having completed cognitive function tests during the initial evaluation.

Exclusion Criteria:

* Having a history of a disease that could affect neurological, psychiatric, or cognitive functions.
* Individuals whose use of glasses, contact lenses, or eye health prevents them from using stroboscopic glasses.
* Having had a head, neck, or serious lower/upper extremity injury within the last 6 months.
* Regular use of any medication (especially medications that affect attention/cognitive functions).
* Individuals who declared they were unable to comply with the study process or who did not participate in follow-up assessments.
* Individuals who did not comply with the research protocol during testing or whose data were incomplete.

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male
Study Population: Adolescent male volleyball players between the ages of 13-18.
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Visual-Spatial Perception | Eight weeks
  Line Orientation Test
Cognitive Functions | Eight weeks
  Trail Making Test
Directing attention | Eight weeks
  Stroop Test

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University of Applied Sciences Physiotherapy and Rehabilitation Research Center, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No